CLINICAL TRIAL: NCT02780830
Title: A Modular Phase I/IIa, Open-Label, Multicentre Study to Assess AZD2014 in Combination With Novel Anti-Cancer Agents in Patients With Relapsed or Refractory Diffuse Large B Cell Lymphoma (INHIBITOR Study)
Brief Title: AZD2014 Plus Novel Anti-Cancer Agents in Relapsed or Refractory Diffuse Large B-Cell Lymphoma
Acronym: INHIBITOR
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study D2276C00001 was not started. No patients were enrolled. The sponsor decided to pursue an alternate design.
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D2276C00001; LYM 103 (Other: Sarah Cannon Research Institute)
Record Dates: First submitted 2016-04-27; First posted 2016-05-24 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-09

CONDITIONS: Core: Relapsed or Refractory Diffuse Large B-Cell Lymphoma; Module 1: Non-GCB Diffuse Large B-Cell Lymphoma
Keywords: Lymphoma; Diffuse Large B-Cell Lymphoma; non-GCB Diffuse Large B-Cell Lymphoma; Relapsed or Refractory non-GCB Diffuse Large B-Cell Lymphoma; Vistusertib; AZD2014; Ibrutinib; Imbruvica
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma; Recurrence | interventions — vistusertib; ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AZD2014 plus Ibrutinib Combination (Experimental): AZD2014 and ibrutinib will be dosed together in the morning under fasting conditions. When possible, the morning doses of AZD2014 and ibrutinib should be taken at approximately the same time each day. The morning doses must be taken in a fasted state (water to drink only) from at least 2 hours prior to the dose to at least 1 hour post dose. AZD2014 will be taken orally twice per day on an intermittent dosing schedule, 2 days on and 5 days off of each week. On days of AZD2014 dosing, ibrutinib will be taken with the morning dose of AZD2014.
  Interventions: Drug: AZD2014; Drug: Ibrutinib

INTERVENTIONS:
Drug: AZD2014 — AZD2014 will be supplied as oral tablets. AZD2014 will be taken orally twice per day on an intermittent dosing schedule, 2 days on and 5 days off of each week.
  Other Names: Vistusertib
Drug: Ibrutinib — Ibrutinib will be provided in hard gelatin capsules in opaque high-density polyethylene bottles. On days of AZD2014 dosing, ibrutinib will be taken with the morning dose of AZD2014.
  Other Names: IMBRUVICA®

SUMMARY:
This is a modular study of AZD2014 in combination with novel anti-cancer agents in patients with different subtypes of relapsed or refractory Diffuse Large B-Cell Lymphoma (DLBCL). Module 1, a combination with ibrutinib in patients with non-germinal centre B-cell-like (non-GCB) DLBCL, will consist of Part A, a Phase I dose-finding arm in which the safety and tolerability of the combination will be assessed, and Part B, a Phase II dose-expansion phase to assess the efficacy of the combination.

DETAILED DESCRIPTION:
This is a modular, Phase I/IIa, open-label, multicentre study of AZD2014, administered orally, in combination with up to 2 novel anti-cancer agents, to patients with different subtypes of relapsed or refractory DLBCL.

Module 1 will assess the combination of AZD2014 and ibrutinib in patients with non-GCB DLBCL and will consist of 2 parts. Part A will be a Phase I dose-finding study in which the safety and tolerability of the combination will be assessed. Part B will be a Phase IIa single-arm dose-expansion phase to assess the efficacy of the combination.

Part A will follow a Continuous Reassessment Method (CRM) based on a Bayesian Adaptive Design to identify the AZD2014/ibrutinib dose combinations where the incidence of dose-limiting toxicity (DLT) is less than 33% during the first cycle. It is anticipated that approximately 30 evaluable patients with non-GCB DLBCL who are not eligible for stem cell transplant may be enrolled. The total number of patients, however, will depend upon the number of cohorts necessary to establish a tolerated combination dose. Determination of tolerated doses will be primarily based on the DLTs seen in Cycle 1. Each cycle will be 28 days. Part A will also include an assessment of single- and multiple-dose pharmacokinetics of the combination of AZD2014 and ibrutinib.

In Part B approximately 50 evaluable patients with non-GCB DLBCL will be enrolled. Patients will receive AZD2014 and ibrutinib at the doses established in Part A in 28-day cycles until there is unacceptable toxicity, disease progression, or the patient withdraws consent. Assessment for response or progressive disease will occur after Cycle 3 and every 3 cycles through the first year, and then every 6 cycles (6 months) thereafter.

In Part B, predictive power monitoring will be used, which could result in stopping Part B for futility. An administrative interim analysis of overall response rate will be conducted thereafter for internal decision making, and the primary analysis will be conducted following data analysis at the primary data cut-off date. The criteria for success will be based on a confidence interval (CI) approach.

Part B will also include an assessment of the impact of repeat intermittent treatment of AZD2014 at the MTD on the pharmacokinetics (PK) of ibrutinib in a sub-group of 9 patients (Part B1). The remaining 41 patients (Part B2) will have sparse PK sampling.

In order to be eligible for Module 1 participants must have pathologically confirmed DLBCL of non-GCB subtype. Participants meeting any of the following criteria may not be enrolled in Module 1:

1. Previous treatment with a Bruton's tyrosine kinase (BTK) inhibitor and/or mammalian target of rapamycin (mTOR) pathway inhibitors.
2. History of severe allergic or anaphylactic reactions to kinase inhibitors or history of hypersensitivity to active or inactive excipients of ibrutinib or drugs with a similar chemical structure or class to ibrutinib.
3. Recent infection requiring systemic treatment that was completed within 14 days prior to the first dose of study drug.

ELIGIBILITY:
Core Inclusion Criteria

1. Males and Females (M/F) ≥18
2. Histopathologically confirmed DLBCL
3. Progressive Disease (PD) after autologous stem cell transplantation (ASCT) or ineligible for ASCT
4. Relapsed/refractory de novo disease, defined as: i) recurrence of disease after complete response (CR), partial response (PR), or stable disease (SD); or ii) PD after completion of previous treatment regimen
5. ≥1 lesion on computerized tomography (CT) or magnetic resonance imaging (MRI) >1.5 cm
6. Adequate hematologic function
7. Adequate hepatic and renal function
8. Prothrombin time (PT)/international normalised ratio (INR) <1.5 x upper limit of normal (ULN) and activated partial thromboplastin time <1.5 x ULN
9. Serum potassium within normal limits (WNL)
10. ECOG perf. status of 0 or 1
11. Female patients willing to use 2 forms of contraception, not breast feeding
12. Male patients surgically sterile or willing to use effective barrier method of contraception

Core Exclusion Criteria

1. Previous allogenic stem cell transplant. Patients may have previous ASCT > 3 months prior
2. Prior standard anti-lymphoma therapy or radiation therapy ≤ 14 days
3. Concurrent systemic immunosuppressive therapy ≤ 28 days
4. Major surgery < 4 weeks or minor surgery < 14 days
5. Haemopoeitic growth factors < 7 days or pegylated G-CSF and darbepoetin < 14 days
6. History of severe allergic or anaphylactic reactions to kinase inhibitors or hypersensitivity to active or inactive excipients of vistusertib
7. Live, attenuated vaccine < 4 weeks
8. Unresolved toxicities from prior anti-cancer therapy with the exception of alopecia.
9. Bleeding disorders or haemophilia
10. History of stroke or intracranial haemorrhage < 6 months
11. Central nervous system (CNS) involvement by lymphoma or spinal cord compression
12. Corticosteroid use with the exception of control of symptoms relating to underlying disease and/or corticosteroid for other indications up to 20 mg/day prednisone
13. History of other malignancies
14. History of HIV, active or chronic hepatitis C, or hepatitis B
15. Have undergone any of the following procedures or experienced conditions currently or < 6 months: coronary artery bypass graft, angioplasty, vascular stent, myocardial infarction, angina pectoris, congestive heart failure [New York Heart Association (NYHA) grade ≥ 2], ventricular arrhythmias requiring continuous therapy, supraventricular arrhythmias, atrial fibrillation, haemorrhagic or thrombotic stroke, TIA or CNS bleeding.
16. Abnormal echo/MUGA at baseline
17. Mean resting QTc >450 msec obtained from 3 ECGs
18. Factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, or family history of sudden unexplained death <40 years-of-age
19. Type I or uncontrolled Type 2 diabetes mellitus.
20. Clinically significant pre-existing renal disease or high risk of developing renal impairment.
21. Refractory nausea and vomiting, malabsorption syndrome, disease significantly affecting GI function, resection of stomach or small bowel, symptomatic inflammatory bowel disease or ulcerative colitis, or partial or complete bowel obstruction.
22. Concomitant use of therapeutic anticoagulants with the exception of short-acting heparins
23. Exposure to potent or moderate inhibitors or inducers of CYP 3A4/5, multi drug resistance 1 (MDR1) permeability glycoprotein (Pgp), or breast cancer resistance protein (BCRP)
24. Exposure to sensitive or narrow therapeutic range substrates of the drug metabolising enzymes CYP2C8, CYP2C9, CYP2C19, CYP2D6 or the drug transporters Pgp (MDR1), BCRP, OATP1B1, OATP1B3, OCT1 and OCT2.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-06; Primary Completion 2019-04 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
The incidence of adverse events (including adverse events detected via laboratory assessment, vital signs and ECG) (Part A). | Throughout the study, approximately 9 months.
  Safety and tolerability will be assessed through the incidence of adverse events. Adverse events will include significant findings on vital signs, clinical chemistry/haematology, coagulation parameters, and electrocardiograms (ECGs).
Overall Response Rate (ORR) in patients with relapsed or refractory DLBCL receiving the combination of AZD2014 and ibrutinib (Part B only) by assessment of the proportion of patients with tumour response. | ORR will be determined at prespecified intervals as the percentage of patients with a documented response before progression or other anti-cancer therapy, assessed up to 5 years.
  ORR will be assessed through the proportion of patients who achieve a disease response (i.e. complete response or partial response) according to the Cheson revised response criteria for malignant lymphoma (2014)
Maximum Tolerated Dose (MTD) | 28 days (1 cycle)
  The safety dose-finding portion of each module (Part A) will follow a Bayesian adaptive design, whereby patients will be enrolled to ensure 3-6 evaluable patients per dose to determine the Recommended Phase 2 Dose (RP2D) and/or MTDs of the combination being studied. The Bayesian Adaptive Design Scheme will utilize a practical Continuous Reassessment Method (CRM) as described in each individual module. Determination of tolerated doses will be primarily based on the DLTs seen in Cycle 1.

SECONDARY OUTCOMES:
The incidence of adverse events (including adverse events detected via laboratory assessment, vital signs and ECG) (Part B). | Throughout the study, approximately 9 months.
  Safety and tolerability will be assessed through the incidence of adverse events. Adverse events will include significant findings on vital signs, clinical chemistry/haematology, coagulation parameters, and ECGs.
Cmax of AZD2014 and ibrutinib following single (Cycle 1 Day 1 Part A, Cycle 0 Day 3 Part B1) and multiple dose. | Single dose and Cycle 1 Day 22
  Plasma pharmacokinetics (PK) - AZD2014 (Part A only) and ibrutinib (Part A and B1) maximum concentration.
AUC for AZD2014 and ibrutinib following single (Cycle 1 Day 1 Part A, Cycle 0 Day 3 Part B1) and multiple dose. | Single dose and Cycle 1 Day 22 over 12 hours (AZD2014) and 24 hours (ibrutinib) post dose
  Plasma PK - AZD2014 (Part A only) and ibrutinib (Part A and B1) area under concentration time curve.
Overall Response Rate (ORR) in patients with relapsed or refractory DLBCL receiving the combination of AZD2014 and ibrutinib (Part A only) by assessment of the proportion of patients with tumour response. | ORR will be determined at prespecified intervals as the percentage of patients with a documented response before progression or other anti-cancer therapy, assessed up to 5 years.
  ORR assessed through the number of patients who achieve a disease response (i.e. complete response or partial response) as assessed by the Cheson revised response criteria for malignant lymphoma (2014).
The anti-tumour activity of the combination of AZD2014 and ibrutinib will be determined in Part A and Part B patients by evaluating duration of response (DoR) by assessment of the amount of time tumour response is maintained. | The DoR will be determined at prespecified intervals from the time of first response to the date of first documented progression, date of death from any cause, or start of other anti-cancer therapy, whichever comes first, assessed up to 5 years.
  DoR will be assessed as the time between disease response being achieved and progressive disease as assessed by the Cheson revised response criteria for malignant lymphoma (2014) or death (in the absence of progression).
The anti-tumour activity of the combination of AZD2014 and ibrutinib will be determined in patients in both Parts A and B by evaluating disease control rate (DCR) at 24 weeks as the percentage of patients who achieve stable disease or a tumour response. | 24 weeks of treatment
  DCR will be assessed through the percentage of patients who achieve stable disease or a disease response (i.e. complete response or partial response) at 24 weeks of treatment without an intervening progression as assessed by the Cheson revised response criteria for malignant lymphoma (2014).
The anti-tumour activity of the combination of AZD2014 and ibrutinib will be determined in Part A and Part B patients by evaluating progression-free survival (PFS). | PFS will be assessed from the date of first dose until the date of first documented progression, date of death from any cause, or start of other anti-cancer therapy, whichever comes first, assessed up to 5 years.
  PFS will be assessed as the time from start of dosing until the date of progression as assessed by the Cheson revised response criteria for malignant lymphoma (2014) or death in the absence of progression.

CONTACTS AND LOCATIONS:
Overall Officials: Ian W Flinn, MD, PhD, Study Chair — SCRI Development Innovations, LLC